CLINICAL TRIAL: NCT00269048
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group, Dose-ranging Study of SB-480848, an Oral Lipoprotein-associated Phospholipase A2 (Lp-PLA2) Inhibitor, in Subjects With Stable Coronary Heart Disease (CHD) or CHD-risk Equivalent to Examine Chronic Inhibition of Lp-PLA2 Effects on Circulating Biomarkers Associated With Cardiovascular Risk, Safety and Tolerability Over 12 Weeks
Brief Title: SB-480848 In Subjects With Coronary Heart Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LPL104884
Record Dates: First submitted 2005-12-21; First posted 2005-12-23 (Estimated); Last update posted 2016-08-08 (Estimated); Status verified 2016-08

CONDITIONS: Atherosclerosis
Keywords: CHD; Lp-PLA2; SB-480848
MeSH Terms: conditions — Atherosclerosis | interventions — darapladib

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): SB-480848
  Interventions: Drug: SB-480848
- Arm 2 (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: SB-480848 — SB-480848
  Arms: Arm 1
Drug: placebo — placebo
  Arms: Arm 2

SUMMARY:
This trial of SB-480848 in approximately 920 subjects with Coronary Heart Disease (CHD) or CHD-risk equivalent will examine whether SB-480848 produces sustained inhibition of plasma Lp-PLA2 activity, explore the effects of SB-480848 on other circulating biomarkers associated with cardiovascular risk, and evaluate the pharmacokinetics, safety and tolerability of SB-480848 over 12 weeks of once-daily oral dosing. Subjects will first be randomized 1:1 to double-blind atorvastatin 20 mg or 80 mg once daily for a minimum of 3 weeks. Subjects will then be randomized 1:1:1:1 to oral doses of SB-480848 40 mg, 80 mg, 160 mg or placebo once daily for 12 weeks. Blood samples will be collected at various timepoints. Vital signs, electrocardiograms, clinical laboratory safety tests and adverse event assessments will be performed to evaluate the safety and tolerability of SB-480848.

DETAILED DESCRIPTION:
A multicenter, randomized, double-blind, placebo-controlled, parallel-group, dose-ranging study of SB-480848, an oral lipoprotein-associated phospholipase A2 (Lp-PLA2) inhibitor, in subjects with stable coronary heart disease (CHD) or CHD-risk equivalent to examine chronic inhibition of Lp-PLA2, effects on circulating biomarkers associated with cardiovascular risk, safety and tolerability over 12 weeks

ELIGIBILITY:
Inclusion criteria:

* Female subjects must be of non-childbearing potential.
* Stable CHD or CHD-risk equivalent.
* Must have been on a stable dose of a statin for =4 weeks with LDL <130 mg/dL (3.4 mmol/L) or off statin therapy for =4 weeks with LDL <160 mg/dL (4.1 mmol/L).
* On a stable dose of at least one oral antiplatelet agent (e.g., aspirin, clopidogrel, or ticlopidine).

Exclusion criteria:

* Recent cardiovascular event and / or vascular procedure.
* History of difficult to manage dyslipidemia.
* Planned cardiac surgery or PCI (percutaneous coronary intervention) or planned major non-cardiac surgery.
* Inadequately controlled hypertension.
* Poorly controlled diabetes mellitus.
* Serum triglycerides >400 mg/dL (4.52 mmol/L).
* Recent or ongoing acute infection.
* History of chronic inflammatory disease.
* Receiving topical, oral, inhaled or injectable corticosteroids.
* History of chronic viral hepatitis, or other chronic hepatic disorders.
* History of kidney transplant.
* History of myopathy or inflammatory muscle disease, or elevated total serum CK (3 x ULN).
* Severe heart failure (NYHA class III or IV), or severe left ventricular dysfunction (ejection fraction <30%).
* Asthma manifested by bronchospasm in the past 6 months, or currently taking inhaled bronchodilator on regular basis.
* History of anaphylaxis, anaphylactoid reactions or severe allergic responses within the past 6 months.
* Malignancy within the past 2 years, other than non-melanoma skin cancer.
* Current life-threatening condition other than vascular disease that may prevent a subject from completing the study.
* QTc interval >440 msec (males) or >450 msec (females).
* Alcohol or drug abuse within the past 6 months.
* Previous exposure to SB-480848.
* Use of an investigational drug within 30 days or 5 half-lives (whichever is the longer) preceding the first dose of study medication (blinded atorvastatin).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 969 (Actual)
Dates: Start 2005-11; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
On treatment sustained inhibition of plasma Lp-PLA2 activity. | 12 Weeks

SECONDARY OUTCOMES:
Difference in dose-dependent effects of SB-480848 on plasma Lp-PLA2 activity, other biomarkers, and safety. | 12 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (99):
- United States (27):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Northport, Alabama
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Spring Valley, California
  - GSK Investigational Site, Torrance, California
  - GSK Investigational Site, Walnut Creek, California
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Pembroke Pines, Florida
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Lacombe, Louisiana
  - GSK Investigational Site, Slidell, Louisiana
  - GSK Investigational Site, Auburn, Maine
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Statesville, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Camp Hill, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Bryan, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, Norfolk, Virginia
  - GSK Investigational Site, Richmond, Virginia
- Argentina (2):
  - GSK Investigational Site, Buenos Aires, Buenos Aires
  - GSK Investigational Site, Buenos Aires
- Australia (3):
  - GSK Investigational Site, Kippa-Ring, Queensland
  - GSK Investigational Site, Caulfield, Victoria
  - GSK Investigational Site, Geelong, Victoria
- Bulgaria (2):
  - GSK Investigational Site, Pleven
  - GSK Investigational Site, Sofia
- Canada (3):
  - GSK Investigational Site, Oakville, Ontario
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Sainte-Foy, Quebec
- GSK Investigational Site, Koebenhavn N, Denmark
- Estonia (2):
  - GSK Investigational Site, Tallinn
  - GSK Investigational Site, Tartu
- France (9):
  - GSK Investigational Site, Anzin
  - GSK Investigational Site, Bron
  - GSK Investigational Site, Créteil
  - GSK Investigational Site, Dommartin-lès-Toul
  - GSK Investigational Site, Gières
  - GSK Investigational Site, Montbrison
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Pessac
  - GSK Investigational Site, Toulouse
- Germany (17):
  - GSK Investigational Site, Kippenheim, Baden-Wurttemberg
  - GSK Investigational Site, Haag, Bavaria
  - GSK Investigational Site, Künzing, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Nuremberg, Bavaria
  - GSK Investigational Site, Rednitzhembach, Bavaria
  - GSK Investigational Site, Hamburg, Hamburg
  - GSK Investigational Site, Schwerin, Mecklenburg-Vorpommern
  - GSK Investigational Site, Bochum, North Rhine-Westphalia
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Goch, North Rhine-Westphalia
  - GSK Investigational Site, Witten, North Rhine-Westphalia
  - GSK Investigational Site, Rhaunen, Rhineland-Palatinate
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Berlin, State of Berlin
- Hungary (4):
  - GSK Investigational Site, Budapest
  - GSK Investigational Site, Debrecen
  - GSK Investigational Site, Szeged
  - GSK Investigational Site, Szolnok
- India (3):
  - GSK Investigational Site, Banglore
  - GSK Investigational Site, Hyderabad
  - GSK Investigational Site, New Delhi
- Netherlands (8):
  - GSK Investigational Site, Den Helder
  - GSK Investigational Site, Ede
  - GSK Investigational Site, Enschede
  - GSK Investigational Site, Haarlem
  - GSK Investigational Site, Hoofddorp
  - GSK Investigational Site, Rotterdam
  - GSK Investigational Site, Sneek
  - GSK Investigational Site, Zeist
- New Zealand (2):
  - GSK Investigational Site, Hamilton
  - GSK Investigational Site, Takapuna
- GSK Investigational Site, Karachi, Pakistan
- Romania (2):
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Târgu Mureş
- Spain (13):
  - GSK Investigational Site, Alicante
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Cáceres
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Móstoles/Madrid
  - GSK Investigational Site, Oviedo
  - GSK Investigational Site, Palma de Mallorca
  - GSK Investigational Site, Quart de Poblet, Valencia
  - GSK Investigational Site, Sant Joan d'Alacant
  - GSK Investigational Site, Santa Coloma de Gramanet/Barcelona
  - GSK Investigational Site, Santiago de Compostela
  - GSK Investigational Site, Santiago de Compostela/La Coruña
  - GSK Investigational Site, Tarrasa, Barcelona

REFERENCES:
- [Derived] Mohler ER 3rd, Ballantyne CM, Davidson MH, Hanefeld M, Ruilope LM, Johnson JL, Zalewski A; Darapladib Investigators. The effect of darapladib on plasma lipoprotein-associated phospholipase A2 activity and cardiovascular biomarkers in patients with stable coronary heart disease or coronary heart disease risk equivalent: the results of a multicenter, randomized, double-blind, placebo-controlled study. J Am Coll Cardiol. 2008 Apr 29;51(17):1632-41. doi: 10.1016/j.jacc.2007.11.079. PMID 18436114
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: LPL104884 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: LPL104884 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: LPL104884 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: LPL104884 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: LPL104884 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: LPL104884 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: LPL104884 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register